CLINICAL TRIAL: NCT00251810
Title: Can CSM Monitor Depth of Anaesthesia Just as Good as BIS?
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: Danmeter (Denmark) (Unknown); The Research Council of Norway (Other)
Responsible Party: Professor MD PhD Johan Rader, Oslo University Hospital
Other Study IDs: CSMtrial
Record Dates: First submitted 2005-11-09; First posted 2005-11-10 (Estimated); Last update posted 2011-08-16 (Estimated); Status verified 2011-08

CONDITIONS: General Anaesthesia
Keywords: general anaesthesia; depth of hypnosis; Cerebral State Monitor; CSM; Bispectral Index; BIS
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- general anaesthesia
  Interventions: Device: Cerebral State Monitor

INTERVENTIONS:
Device: Cerebral State Monitor — All patients monitored with BIS and CSM, results hidden for the anesthesiologist.

SUMMARY:
This study aims to test whether two depth-of-anaesthesia-monitors can perform equally well in monitoring anaesthetic sleep, both at induction and emergence from anaesthesia and during surgery.

DETAILED DESCRIPTION:
There is a considerable variation in the need of anaesthetics for the individual patient. For measuring the hypnotic component (i.e. sleep) during anaesthesia, no reliable monitoring system was available before Bispectral Index, BIS (Aspect Medical) was commercially launched about ten years ago. BIS is based on complex mathematical and statistical processing of the electroencephalogram, EEG.

A widespread use of BIS has been limited in part by high costs. Last year a considerably cheaper EEG monitor, Cerebral State Monitor, CSM (Danmeter), was launched into the marked. The validation of CSM is so far limited to very few cases comparing BIS and CSM offline. No large scaled clinical study has been performed to test whether CSM also reflects depth of hypnosis in a reliable way.

We set up a study on 60 relatively healthy patients, undergoing various kind of surgery in general anaesthesia. The study is approved by the Regional Committee of Ethics in Medicine, Health Region East, and all patients give written informed consent. Both monitors (BIS and CSM) are applied to the patients, but only information from BIS is available for the anaesthetist throughout surgery. Information from the two monitors and from the routine monitoring equipment as well as from the actual delivery of anaesthetics is sampled online into a designed data program (Rugloop, Demed, Belgium).

The output from BIS and CSM will afterwards be analyzed together with statistical experts, to see if CSM can predict the time for falling asleep and time for awakening just as good as BIS. The curves for the two monitors will also be compared, qualitatively and quantitatively, to see if they perform equally well.

Inclusion criterias:

* Written informed consent
* ASA 1-3
* Age 18 - 75
* Surgery in all parts of the body except from the face/head in general anaesthesia; surgery expected to last for 30 - 120 minutes

Exclusion criterias:

* Extreme over- or underweight
* Epilepsy or other conditions or medications that would probably influence on the EEG
* Alcohol- or drug abuse
* Contraindication for the actual anaesthetics, being propofol and remifentanil

ELIGIBILITY:
Inclusion Criteria:

* Healthy patients undergoing surgery in general anaesthesia

Exclusion Criteria:

* No ability to give written informed consent, drug abuse, patients on medication suspected or known to influence the EEG, surgery involving head or face

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 60 patients undergoing general anaesthesia
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2004-11

CONTACTS AND LOCATIONS:
Overall Officials: Johan Raeder, professor, Study Chair — University of Oslo
Locations (1):
- Department of Anaesthesia, Ullevaal University Hospital, Oslo, Norway